CLINICAL TRIAL: NCT02830100
Title: Neural Correlates of Intern Speech
Acronym: INNERSPEECH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no more subjects for recrutment
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC14.304
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteer
Keywords: Intern speech; Speech and visual imaging; Mind and oral drift; Cognitive performance; Magnetic Resonance Imaging
MeSH Terms: conditions — Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Other)
  Interventions: Other: Healthy volunteers; Device: MRI

INTERVENTIONS:
Other: Healthy volunteers — Magnetic Resonance Imaging during intern speech, listening, talking, thinking.
Device: MRI

SUMMARY:
The goal is to define what is the nature of intern speech, how it manifests itself, who deal with agency in intern speech and finally what is the role of intern speech in attention tasks.

DETAILED DESCRIPTION:
Intern speech has a main goal in memory, thinking and self-awareness. So this study might bring information in order to better understand any potential adverse effect on depression or anxiety disorders for example.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years
* Right-handed
* French as mother tongue
* Visual acuity that allow to read stimulis (contact lens authorized)
* Healthy subject

Exclusion Criteria:

* Respiratory or cardio-vascular pathology
* Claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2015-12-12 (Actual); Study Completion 2015-12-12 (Actual)

PRIMARY OUTCOMES:
Study intern speech | About an hour
  Magnetic Resonance Imaging while talking, thinking, listening

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Krainik, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Baciu MV, Rubin C, Decorps MA, Segebarth CM. fMRI assessment of hemispheric language dominance using a simple inner speech paradigm. NMR Biomed. 1999 Aug;12(5):293-8. doi: 10.1002/(sici)1099-1492(199908)12:53.0.co;2-6. PMID 10484818
- [Background] Basho S, Palmer ED, Rubio MA, Wulfeck B, Muller RA. Effects of generation mode in fMRI adaptations of semantic fluency: paced production and overt speech. Neuropsychologia. 2007 Apr 9;45(8):1697-706. doi: 10.1016/j.neuropsychologia.2007.01.007. Epub 2007 Jan 16. PMID 17292926
- [Background] Bookheimer SY, Zeffiro TA, Blaxton T, Gaillard W, Theodore W. Regional cerebral blood flow during object naming and word reading. Human Brain Mapping. 1995;3:93-106.
- [Background] Clark A, Karmiloff-Smith A. The cognizer's innards: a psychological and philosophical perspective on the development of thought. Mind & Language. 1993;8:487-519.
- [Background] Conrad B, Schonle P. Speech and respiration. Arch Psychiatr Nervenkr (1970). 1979 Apr 12;226(4):251-68. doi: 10.1007/BF00342238. PMID 454139
- [Background] Davis RN, Nolen-Hoeksema S. Cognitive inflexibility among ruminators and nonruminators. Cognitive Therapy and Research. 2000;24:699-711.
- [Background] Frings M, Dimitrova A, Schorn CF, Elles HG, Hein-Kropp C, Gizewski ER, Diener HC, Timmann D. Cerebellar involvement in verb generation: an fMRI study. Neurosci Lett. 2006 Nov 27;409(1):19-23. doi: 10.1016/j.neulet.2006.08.058. Epub 2006 Oct 12. PMID 17046160
- [Background] Huang J, Carr TH, Cao Y. Comparing cortical activations for silent and overt speech using event-related fMRI. Hum Brain Mapp. 2002 Jan;15(1):39-53. doi: 10.1002/hbm.1060. PMID 11747099
- [Background] Lupyan G. Extracommunicative functions of language: verbal interference causes selective categorization impairments. Psychon Bull Rev. 2009 Aug;16(4):711-8. doi: 10.3758/PBR.16.4.711. PMID 19648457
- [Background] McGuire PK, Silbersweig DA, Murray RM, David AS, Frackowiak RS, Frith CD. Functional anatomy of inner speech and auditory verbal imagery. Psychol Med. 1996 Jan;26(1):29-38. doi: 10.1017/s0033291700033699. PMID 8643761
- [Background] Morin A. Inner Speech Encyclopedia of Human Behavior. 2012;Elsevier:436-43.
- [Background] Netsell R, Ashley E, Bakker K. The Inner Speech of Persons who Stutter. Proceedings of the International Motor Speech Conference. Savannah, Georgia2010
- [Background] Olivers CN, Nieuwenhuis S. The beneficial effects of additional task load, positive affect, and instruction on the attentional blink. J Exp Psychol Hum Percept Perform. 2006 Apr;32(2):364-79. doi: 10.1037/0096-1523.32.2.364. PMID 16634676
- [Background] Owen WJ, Borowsky R, Sarty GE. FMRI of two measures of phonological processing in visual word recognition: ecological validity matters. Brain Lang. 2004 Jul-Sep;90(1-3):40-6. doi: 10.1016/S0093-934X(03)00418-8. PMID 15172523
- [Background] Palmer ED, Rosen HJ, Ojemann JG, Buckner RL, Kelley WM, Petersen SE. An event-related fMRI study of overt and covert word stem completion. Neuroimage. 2001 Jul;14(1 Pt 1):182-93. doi: 10.1006/nimg.2001.0779. PMID 11525327
- [Background] Partovi S, Konrad F, Karimi S, Rengier F, Lyo JK, Zipp L, Nennig E, Stippich C. Effects of covert and overt paradigms in clinical language fMRI. Acad Radiol. 2012 May;19(5):518-25. doi: 10.1016/j.acra.2011.12.017. Epub 2012 Jan 27. PMID 22281389
- [Background] Rosen HJ, Ojemann JG, Ollinger JM, Petersen SE. Comparison of brain activation during word retrieval done silently and aloud using fMRI. Brain Cogn. 2000 Mar;42(2):201-17. doi: 10.1006/brcg.1999.1100. PMID 10744920
- [Background] Shergill SS, Bullmore ET, Brammer MJ, Williams SC, Murray RM, McGuire PK. A functional study of auditory verbal imagery. Psychol Med. 2001 Feb;31(2):241-53. doi: 10.1017/s003329170100335x. PMID 11232912
- [Background] Shuster LI, Lemieux SK. An fMRI investigation of covertly and overtly produced mono- and multisyllabic words. Brain Lang. 2005 Apr;93(1):20-31. doi: 10.1016/j.bandl.2004.07.007. PMID 15766765
- [Background] Uttl B, Morin A, Faulds TJ, Hall T, Wilson JM. Sampling Inner Speech Using Text Messaging. Proceedings of the Canadian Society for Brain, Behavior, and Cognitive Science. Kingston2012. p. 287.
- [Derived] Roger E, Rodrigues De Almeida L, Loevenbruck H, Perrone-Bertolotti M, Cousin E, Schwartz JL, Perrier P, Dohen M, Vilain A, Baraduc P, Achard S, Baciu M. Unraveling the functional attributes of the language connectome: crucial subnetworks, flexibility and variability. Neuroimage. 2022 Nov;263:119672. doi: 10.1016/j.neuroimage.2022.119672. Epub 2022 Oct 6. PMID 36209795